CLINICAL TRIAL: NCT03210012
Title: Bubbles, Stress, Diastole
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinica ARS Medica (Other)
Responsible Party: Principal Investigator, Dr. med. Claudio Camponovo, Principal Investigator, Clinica ARS Medica
Other Study IDs: CMAS1
Record Dates: First submitted 2017-06-28; First posted 2017-07-06 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Diastolic Dysfunction; Endothelial Dysfunction
MeSH Terms: interventions — Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for microparticles count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Three dives with different gas mixture : AIR (21% di O2 e 79% di N2), NITROX 32 (32% di O2 e 68% di N2) and TRIMIX (21% O2, 44% N2 e 35% He)
  Interventions: Diagnostic Test: Transthoracic echocardiography; Diagnostic Test: Blood samples

INTERVENTIONS:
Diagnostic Test: Transthoracic echocardiography — Diagnostic test done prior and after the dive
Diagnostic Test: Blood samples — Diagnostic test done prior and after the dive

SUMMARY:
This is a monocentric pilot study to assess the safety profile of a 30-meter deep underwater diving using 3 different type of gas mixtures: AIR (21% O2 and 79% N2), NITROX 32 (32% O2 And 68% N2) and TRIMIX (21% O2, 44% N2 and 35% He).

DETAILED DESCRIPTION:
The participants will be measured for vital parameters, blood samples and transthoracic cardiac ultrasound before diving (baseline).

Participants will be requested to perform recreational dive, which does not require particular decompression stops, at a depth of 30 meters with a 30 minutes botton time. 20 minutes after dive the same measurements as baseline will be repeated, once at rest and once after a physical effort by performing a series of 10 bending on the legs (squats). The day after dive, the participants will be interviewed by phone (FOLLOW-UP) by a physician. It will be required to report any unusual event, MDD symptom, or neurological complication.

Same procedure will be repeated with three different type of blends (AIR, NITROX, TRIMIX).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 60
* healthy subjects
* body mass BMI < a 30
* physical status ASA 1

Exclusion Criteria:

* subjects with significant clinical impairments such as important head trauma, general pain, low back pain, diabetes, asthma, cardiac and coagulation dysfunctions
* pregnant women
* participation in another study in the last 3 months
* use of drugs and alcohol
* smoking
* psychiatric disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healty volunteer divers
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2017-06-11 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Best gas mixture | 1 month
  Best gas mixture with minimal cardiac function impact (endothelial stress)

SECONDARY OUTCOMES:
diastolic function evaluation | 1 month
  diastolic function evaluated after a dive with three different gas mixtures

CONTACTS AND LOCATIONS:
Locations (1):
- Salvataggio Sub Gambarogno, San Nazzaro, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided